CLINICAL TRIAL: NCT01378182
Title: Efficacy of Invitro Expanded Bone Marrow Derived Allogeneic Mesenchymal Stem Cell Transplantation Via Portal Vein or Hepatic Artery or Peripheral Vein in Patients With Wilson Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murat Kantarcioglu (Other)
Collaborators: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Sponsor-Investigator, Murat Kantarcioglu, Gulhane Military Medical Academy, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Organization: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110S153
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Wilson's Disease
Keywords: Transplantation,Stem Cell; Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: allogeneic mesenchymal stem cell transplantation — 1.000.000(one million) cells/kg, IV (1/2 of dose in the Peripheral vein and 1/2 of dose into the right hepatic artery)

SUMMARY:
Wilson's disease is an autosomal recessive genetically inherited disorder of copper metabolism, causing neurological, psychiatric and liver disease. The ATP7B gene on the 13th chromosome is responsible for the disease. Liver has a critical role on copper metabolism. It is the main site of copper accumulation and bile secretion is the only physiologic way of copper elimination. Due to defective production of ceruloplasmin which carries copper, wide amount of free copper precipitates throughout the body but particularly in the liver, eyes and brain. Patients are bound to lifelong chelating agents such as penicillamine, trientine and tetramine dihydrochloride. Unfortunately, these medications may cause severe side-effects such as hypersensitivity reactions, bone marrow suppression, auto-immune disease and sideroblastic anemia. Medical treatment of liver cirrhosis, the last stage of the illness that leads to morbidity and mortality in the Wilson Disease, is difficult. Liver transplantation is still the most effective treatment for the patients with liver cirrhosis in Wilson Disease. However, serious problems are accompanied with liver transplantation. Lack of liver donors, complications during and after the surgery, graft rejection and high costs are the main problems.

There are cells in the human body that are capable to renew themselves and differentiate to a diverse range of specialized cell types. These are called "stem cells". Stem cells can be differentiated to specialized cells in appropriate medias in the laboratory. Recently, the differentiation potential of mesenchymal stem cells into hepatocytes is proved by demonstrating hepatocytes containing Y chromosome in the female who has had bone marrow transplantation from male donors. In many laboratory studies, it is observed that human bone marrow derived mesenchymal stem cells, transplanted to animals with induced liver damage, differentiate into the albumin producing hepatocytes without fusion. By these studies, it is understood that mesenchymal stem cells are more potent than other bone marrow elements in context of differentiation to hepatocytes. Even though the number of studies on human for the same purpose is few, findings are supporting those of animal experiments. Mesenchymal stem cells are non-immunogenic. Safety and feasibility of allogeneic transplantations between individuals without need of immunosuppressive drug regimen are proven. Proofs of correcting metabolic defects by this way are also presented in some publications. For the reasons mentioned above, allogeneic mesenchymal stem cell transplantation is a promising treatment modality especially for the hereditary metabolic diseases. By this way, non-immunogeneic mesenchymal stem cells which have healthy genetic structure, can manufacture the required enzyme, will be repopulated in the damaged tissue and contribute to the clinical improvement.

In this study, mesenchymal stem cells will be derived from healthy volunteer donor's bone marrow and be expanded in-vitro, and then 1 million cells per kg will be infused to patients with liver cirrhosis related to Wilson disease, 50 million cells via hepatic artery and the remaining cells via peripheral vein. It is aimed to enable liver regeneration, decrease fibrosis rate, improve patient's health conditions, increase ceruloplasmin synthesis, ameliorate disorder of copper metabolism, decrease the need for chelating agents, increase living standards of patients, and prolong waiting time for liver transplantation. Finally it is aimed to establish a new and regenerative treatment protocol alternative to liver transplantation. For observation of clinical and laboratory improvement, patients are planned to be monitored by histopathologic examination of liver biopsies before and at 6th month after the treatment, monthly biochemical and hematologic blood tests and periodic radiologic examinations. This is a hopeful, avant garde and sophisticated study which may constitute new horizons in context of cellular therapies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical, radiologic and pathologically proven Wilson's Disease with hepatic presentation
* Patients with no hepatic malignancies
* No co-existing serious respiratory and/or cardiovascular morbidities
* Patients who approved to join the study group with informed and written consent
* Patients with platelet count more than 30.000/mm3

Exclusion Criteria:

* Clinical diagnosis of Wilson's Disease with neuropsychiatric presentation
* Current alcohol consumption
* Patients who have acute or chronic viral hepatitis infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
differantiation of transplanted mesenchymal stem cells to hepatocytes in post treatment liver biopsies | liver biopsies performed at sixth month after mesenchymal stem cell transplantation
  all patients will be transplanted bone marrow derived mesenchymal stem cells belonging to the opposite sex in order to genetically determine the mature hepatocyte

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology; Gulhane Military Medical Academy, Ankara, Turkey (Türkiye)